CLINICAL TRIAL: NCT02515188
Title: The Effect of Additional Propacetamol Infusion on Post Procedural Outcome and Opioid Consumption During Catheter Ablation of Atrial Fibrillation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2015-0502
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — propacetamol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- propacetamol group (Experimental)
  Interventions: Drug: Propacetamol
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propacetamol — Randomly selected patients of the propacetamol group are given intravenous propacetamol 2g for 15 minutes on the beginning of the procedure.
  Other Names: Propacetamol (Denogan®, Yungjin, Seoul, Korea)
  Arms: propacetamol group
Drug: Placebo — Placebo group are given intravenous Normal Saline 2g for 15 minutes on the beginning of the procedure.
  Other Names: Normal Saline
  Arms: placebo group

SUMMARY:
Sedation for catheter ablation of atrial fibrillation should be performed to achieve analgesia, immobilization, and maintenance of airway. Various anesthetic agents such as propofol, dexmedetomidine, and midazolam were investigated to achieve this goal. However, propofol and midazolam causes respiratory depression and dexmedetomidine occasionally accompanies hypotension or hypertension and bradycardia. Therefore, anesthetic agent that does not induce respiratory depression with stable hemodynamics is needed.

Propacetamol (Denogan®, Yungjin, Seoul, Korea) is injectable prodrug of acetaminophen and 1st line drug for fever and pain. In a previous study, paracetamol reduced morphine consumption after surgery. And paracetamol does not cause respiratory depression. Thus, the investigators hypothesized that addition of propacetamol to previously used sedatives midazolam-remifentanil will reduce opioid consumption during the catheter ablation.

Therefore, the investigators designed this study to investigate the role of addition of propacetamol to previous used midazolam-remifentanil sedation. This study will compare the opioid consumption and respiratory effect of propacetamol with placebo-control for catheter ablation of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo catheter ablation for arrhythmia

Exclusion Criteria:

* Subjects are ineligible if they have liver disease, kidney disease,
* American society of anesthesiology class 3 or 4,
* age under 20 years,
* cognitive dysfunction,
* disabling mental change disorder,
* patients are unable to communicate or speak Korean

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-06-23 (Actual)

PRIMARY OUTCOMES:
total amount of opioid consumption | 1 day
  Total opioid consumption during the procedure will be recorded. And post procedural consumption of analgesics also will be recorded.

SECONDARY OUTCOMES:
Respiratory rate | 1 day
Depth of sedation | 1 day
  depth of sedation measured by Ramsay Sedation Score
Post procedural pain | 1 day
  post procedural pain measured by consumption of analgesics and VAS (Visual Analog Scale)
nausea point | 1 day
  nausea measured by 11-point NRS (Numerical Rating Scale)
number of vomiting | 1 day
intra-procedural hemodynamics | 1 day
  intra-procedural hemodynamics measured by amount of used vasopressors
satisfaction of patients | 1 day
  satisfaction of patient and surgeons measured by 5-point NRS
recovery time | 1 day
  monitored with heart rate and blood pressure
satisfaction of surgeons | 1 day
  satisfaction of patient and surgeons measured by 5-point NRS

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea